CLINICAL TRIAL: NCT05315076
Title: Comparison of Thoracic Manipulation and Muscle Energy Technique in Non-specific Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC 01211 Muhammad Saad Hassan
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Neck Pain
Keywords: Pain; thoracic manipulation; muscle energy technique; disability; range of motion
MeSH Terms: conditions — Neck Pain; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracic Manipulation Posterior anterior and conventional therapy (Experimental): Thoracic Manipulation Posterior anterior and conventional therapy
  Interventions: Other: thoracic Manipulation Posterior anterior and conventional therapy; Other: Muscle Energy Technique (PIR) and conventional treatment
- Muscle Energy Technique (PIR) and conventional treatment (Experimental): Muscle Energy Technique (PIR) and conventional treatment
  Interventions: Other: thoracic Manipulation Posterior anterior and conventional therapy; Other: Muscle Energy Technique (PIR) and conventional treatment

INTERVENTIONS:
Other: thoracic Manipulation Posterior anterior and conventional therapy — A high-velocity, end range force directed to both sides of the respective zygapophyseal joint as indicated by the segmental examination. This procedure will be performed for a maximum of two attempts. When a cracking sound occurred, the therapist will move on to the next segmental restriction from an upper level to a lower level.
Other: Muscle Energy Technique (PIR) and conventional treatment — sustain the Isometric contraction for 7-10 and hold the breath. Then the patient will be asked to breathe out and relax while the therapist stretches further up to the neck barrier and hold this for 30 seconds.3 to 5 repetition

SUMMARY:
To compare the effects of Thoracic manipulation and MET in relieving pain.in improving Range of motion and in improving functional disability.

DETAILED DESCRIPTION:
Neck pain is a common musculoskeletal disorder. Mechanical neck pain is also known as non-specific neck pain and is defined as the pain anywhere within the region bounded superiorly by superior nuchal line, inferiorly by an imaginary line through the tip of first thoracic spinous process and laterally by sagittal plane tangential to the lateral borders of the neck in which pain is provoked by sustained neck posture, neck movement, pain on palpation of cervical musculature without pathologies. In most patients, neck pain can be a common cause of disability: it is associated with daily activity limitations, reduction of work productivity and decrease in quality of life. Mechanical neck pain is commonly seen in people involved in occupation like computer processing, clerical job, students and people with sedentary life style awkward occupational posture, heavy lifting and physically demanding work.

thoracic spine manipulation (TSM) is defined as a high-velocity/low amplitude movement or "thrust" directed at any segment of the thoracic spine.

Muscle energy technique (MET) is a method of treatment that involves the voluntary contraction of subject's muscles in a precisely controlled direction, against a counterforce and producing post isometric relaxation through the influence of the Golgi tendon. MET is used to decrease pain, stretch tight structures muscle and fascia, reduce muscle tone, improve local circulation, and mobilize joint restriction

ELIGIBILITY:
Inclusion Criteria:

* Patients who present with a primary complaint of mechanical neck pain (defined as pain in the region between the superior nuchal line and first thoracic spinous process) with limited Range of motion.
* Patients with non-radiating neck pain of moderate intensity scoring 4-8 on the numeric pain rating scale (NPRS).
* Subacute or chronic cases (4 -12 weeks)
* Have a Neck Disability Index (NDI) score of 20% or greater (10 points or greater on a 0-to-50 scale)
* Dull aching neck pain increased by sustained postures, neck movement

Exclusion Criteria:

* Patients with a positive history of trauma, fracture or surgery of the cervical spine.
* Neck pain with radiation to the arm and upper extremity
* Diagnosed cases of torticollis, and scoliosis
* History of osteoporosis, Any heart disease
* Taken previous physiotherapy session.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-05 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | three weeks
  The Numeric Pain Rating Scale (NPRS) measures the subjective intensity of pain. The NPRS is an eleven-point scale from 0 to 10. "0" = no pain and "10" = the most intense pain imaginable.Assesment to be done at baseline,1st session,3rd session and 6th session.
Inclinometer | three weeks
  it is used for measurements of cervical flexion, extension, lateral flexion, and rotation.Assesment to be done at baseline,1st session,3rd session and 6th session.
Neck Disability Index | three weeks
  The neck disability index is a ten-item self-reported questionnaire that assesses pain and associated disability, with a total max score of 50 points. .Assessment to be done at baseline,1st session,3rd session and 6th session.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Khalid, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Rawal dental and general hospital,, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No